CLINICAL TRIAL: NCT05773677
Title: FIT: Food in Twins. Diet in Twin Pregnancy: the Wellness of Mother and Babies.
Brief Title: Diet in Twin Pregnancy: the Wellness of Mother and Babies.
Acronym: FIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Visconti Daniela, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5078
Record Dates: First submitted 2023-02-24; First posted 2023-03-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication; Gestational Diabetes; Gestational Hypertension; Intrahepatic Cholestasis of Pregnancy; Food Habits; Diet, Healthy
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Intrahepatic Cholestasis of Pregnancy; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Case group: prospective Control group: retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group: with diet (Experimental): Prescription of specific diet in pregnancy
  Interventions: Dietary Supplement: Specific Diet
- Control Group: no diet (No Intervention): Retrospective group with no diet

INTERVENTIONS:
Dietary Supplement: Specific Diet — A specific diet will be developed for each patient, which will also take into account any food allergies or intolerances.
  Each diet will be then eventually modified and revised throughout the pregnancy, according to the evolution of the same.
  Arms: Case Group: with diet

SUMMARY:
The aim of this study is to evaluate how variations in maternal nutrition may affect twin pregnancy and in particular:

* incidence of maternal obstetric complications:

  * gestational diabetes
  * gestational hypertension or preeclampsia
  * intrahepatic cholestasis (ICP)
* fetal growth, development and birth weight of the babies

DETAILED DESCRIPTION:
Study design

At the time of recruitment, each patient will perform an initial clinical nutrition examination, during which will be evaluated, on the basis of BMI and specific anthropometric parameters, the necessary nutritional intake.

Patients included in the study will then be classified, on the basis of pre-pregnancy BMI, into 2 classes:

* normal weight (BMI 18-25)
* overweight (BMI 25-30) A specific diet will be developed for each patient, which will also take into account any food allergies or intolerances.

Each diet will be then eventually modified and revised throughout the pregnancy, according to the evolution of the same.

Patients will then continue their regular obstetrical examinations at the Obstetrical Day Hospital, every 4 weeks in case of uncomplicated dichorionic twin pregnancy and every 2 weeks in case of uncomplicated monochorionic twin pregnancy.

Once a month, in coincidence with the appointment at the Obstetric Day Hospital, the enrolled patients will be evaluated by the dedicated team of nutritionists.

ELIGIBILITY:
Inclusion Criteria:

* dichorionic-diamniotic twin pregnancies
* monochorionic-diamniotic twin pregrancies
* monochorionic- monoamniotic twin pregnancies
* spontaneous onset or by homologous PMA techniques
* Age between 18 and 40 years
* Gestational age between 8 weeks+0 days and 25 weeks+6 days

Exclusion Criteria:

* Pregestational diabetes mellitus (type I and II)
* Chronic hypertension
* Previous bariatric surgery
* Chronic gastrointestinal disease (Celiac disease, Crohn's disease, Ulcerative Rectocolitis)
* Age less than 18 years or more than 40 years
* Gestational age less than 8 weeks or more than 26 weeks
* Fetal structural and/or genetic abnormalities
* Heterologous PMA
* Maternal eating disorders
* Drug and/or alcohol use
* Multiple pregnancies with more than two babies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
incidence of maternal obstetric complications: | From enrollment in the study to delivery
  * gestational diabetes
  * gestational hypertension or preeclampsia -intrahepatic cholestasis (ICP)

SECONDARY OUTCOMES:
fetal growth and birth weight of the babies | From enrollment in the study to delivery
  estimated fetal weight and actual fetal weight at delivery (expressed in grams)
maternal weight gain | From enrollment in the study to delivery
  expressed in kilograms
differences in early or late enrollment of patients | From enrollment in the study to delivery
  advantage of early enrollment in reducing the incidence of the above complications (expressed as percentage)

CONTACTS AND LOCATIONS:
Locations (1):
- FPGemelliIRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No